CLINICAL TRIAL: NCT06639854
Title: The Use of Cytomegalovirus Cell Mediated Immunity to Optimize the Duration of Letermovir Prophylaxis in Hematopoietic Cell Transplant Recipients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-1144; NCI-2024-08626 (Other: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Cytomegalovirus Cell Mediated Immunity; Hematopoietic Cell Transplant
MeSH Terms: interventions — letermovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interrupted letermovir prophylaxis (Experimental): Participants assigned to the investigational group, you will also receive letermovir at first, but depending on the result of the study blood tests, your dose may be paused as long as your immune system shows an immune response against CMV.
  Interventions: Procedure: Hematopoietic Cell Transplant; Drug: Letermovir
- Standard letermovir prophylaxis (Experimental): Participants assigned to the standard care group, you will receive treatment with letermovir every day to prevent CMV infection.
  Interventions: Procedure: Hematopoietic Cell Transplant; Drug: Letermovir

INTERVENTIONS:
Procedure: Hematopoietic Cell Transplant — Participants choices may include to receive standard post-transplant virus prevention with letermovir or other standard drugs without being part of this study. Participants may choose to receive other investigational therapy, if available.
  These alternative treatments have risks and benefits that may be the same or different than those in this research study.
Drug: Letermovir — Given by PO

SUMMARY:
The goal of this laboratory research study is to learn if interrupting a patient's letermovir dosing based on their immune system response can help HSC transplant patients avoid post-treatment CMV infections better than taking letermovir every day without interruption.

DETAILED DESCRIPTION:
Primary Objective

•To compare the proportion of CS-CMVi in allo-HCT recipients who had interrupted letermovir prophylaxis based on CMV CMI or extended duration of letermovir prophylaxis up to 200 days post transplantation.

Secondary Objectives

* To compare the proportion of CS-CMVi in HCT recipients who had interrupted letermovir prophylaxis based on CMV CMI or extended duration of letermovir prophylaxis at 365 days post transplantation.
* To compare the overall use of letermovir in HCT recipients in both arms.
* To compare CMV CMI in HCT recipients in both arms.
* To compare all-cause mortality and nonrelapse mortality between the 2 arms at day +200 and day +365.
* Healthcare expenditures for letermovir use and TCIP for both arms from day +100 to day +200.

ELIGIBILITY:
Inclusion criteria

1. Allogeneic HCT recipients with positive CMV serostatus
2. On letermovir prophylaxis at day 90 post transplant (+/- 7 days)
3. At high risk for CMV reactivation after day +100:

   1. Prior or active graft versus host disease requiring systemic steroids
   2. Mismatch stem cell donor (includes haploidentical, mismatch unrelated donor (MMUD), match related donor with at least one mismatch at one of the three specified HLA gene loci (HLA-A, HLA-B, or HLA-DR) and cord donor recipients)
   3. Received T cell depletion or anti thymoglobulin during conditioning
   4. CMV reactivation prior to day 100 post transplant
   5. On steroids at any dose within 2 weeks of enrollment

Exclusion criteria

1. Patients under the age of 18
2. Patients are discharged from our institution and unwilling to come back for follow up
3. Patients are actively undergoing treatment for CS-CMVi at time of screening. Prior CS-CMVi is not an exclusion from study.
4. Patients are allergic or intolerant to letermovir or have history of letermovir resistant CMV infection.
5. Not able to procure letermovir for extended prophylaxis beyond day +100.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs). | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Fareed Khawaja, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org